CLINICAL TRIAL: NCT01618032
Title: The Effects of Two Techniques of Mobilization in the Improvement of Dorsiflexion on Chronic Instability Ankles. A Double Blind Randomized Controlled Trial
Brief Title: Effects of Two Techniques of Mobilization in the Dorsiflexion on Patients With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Principal Investigator, Angel Luis Rodriguez, Professor at Physical Therapy Department, CEU San Pablo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEU-002
Record Dates: First submitted 2012-06-08; First posted 2012-06-13 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Instability of Joint

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HVLA (Experimental): High velocity and low amplitude traction manipulation on the ankle joint
  Interventions: Other: HVLA
- MWM (Experimental): Mobilization with movement on ankle joint as Mulligan
  Interventions: Other: MWM
- placebo (Sham Comparator): Contact without therapeutic effect
  Interventions: Other: placebo

INTERVENTIONS:
Other: HVLA — High velocity and low amplitude manipulation in traction of subtalar jonit
  Arms: HVLA
Other: MWM — Mobilization with movement as Mulligan for increase dorsiflexion of the ankle in weight bearing
  Arms: MWM
Other: placebo — Manual contact during a period of time similar of teh other interventions
  Arms: placebo

SUMMARY:
Restrictions on ankle dorsiflexion are common in subjects with chronic ankle instability (CAI). In fact, this is one factor that can contribute to the recurrence of such injuries. Passive mobilization techniques to improve ankle dorsiflexion are commonly used in physiotherapy treatments. However, no studies have compared manipulative techniques of mobilization techniques in subjects with chronic ankle instability.

The aim of this study is to compare the effects of two mobilization techniques on ankle dorsiflexion in patients with chronic ankle instability.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic ankle instability

Exclusion Criteria:

* Acute or subacute ankle sprain.
* Recent lesions in lower extremities.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pre-intervention ankle dorsiflexion | pre-intervention
  Ankle dorsiflexion is measured by the weight-bearing lunge method
Inmediately post-intervention ankle dorsiflexion | inmediately post-intervention
  Ankle dorsiflexion is measured by the weight-bearing lunge method
ten minutes post-intervention ankle dorsiflexion | ten minutes post-intervention
  Ankle dorsiflexion is measured by the weight-bearing lunge method
24 hr post-intervention ankle dorsiflexion | 24 hr post-intervention
  Ankle dorsiflexion is measured by the weight-bearing lunge method
48 hr post-intervention ankle dorsiflexion | 48 hr post-intervention
  Ankle dorsiflexion is measured by the weight-bearing lunge method

CONTACTS AND LOCATIONS:
Overall Officials: Ángel L Rodríguez-Fernández, PT, MSc, Principal Investigator — CEU San Pablo University; David Marrón-Gómez, PT, MSc, Study Chair — CEU San Pablo University